CLINICAL TRIAL: NCT04054518
Title: Durvalumab (MEDI4736) as Maintenance Treatment Following Chemoradiation for Locally Advanced Unresectable Esophageal Squamous Cell Carcinoma (DESC).
Brief Title: Durvalumab as Maintenance Following Chemoradiation for Unresectable Esophageal Squamous Cell Carcinoma
Acronym: DESC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tiago Biachi (Other)
Responsible Party: Sponsor-Investigator, Tiago Biachi, Principal Investigator, Instituto do Cancer do Estado de São Paulo
Organization: Instituto do Cancer do Estado de São Paulo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1473/19
Record Dates: First submitted 2019-08-08; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Durvalumab (Experimental): 1500 mg durvalumab (MEDI4736) via IV infusion Q4W <<for up to a maximum of 12 months (up to 13 doses/cycles) with the last administration on week 48>> or <<until confirmed disease progression>> unless there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab (MEDI4736) will be supplied as a 500-mg vial solution for infusion after dilution.
  Other Names: MEDI4736

SUMMARY:
Single arm phase II trial designed to assess the efficacy of durvalumab treatment in terms of 6-month progression-free survival. We will include 22 patients who will receive 1500 mg durvalumab (MEDI4736) via IV infusion Q4W <<for up to a maximum of 12 months (up to 13 doses/cycles) with the last administration on week 48>> or <<until confirmed disease progression>> unless there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met. If a patient's weight falls to 30 kg or below for 1 week or longer ( ≥ 7 days) durvalumab will be permanently discontinued.

DETAILED DESCRIPTION:
A) Study Title: Durvalumab (MEDI4736) as maintenance treatment following chemoradiation for locally advanced unresectable esophageal squamous cell carcinoma (DESC)

B) Protocol Number: ESR-17-12757

C) Clinical Phase: 2

D) Study Duration: 36 months

E) Investigational Product(s) and Reference Therapy: Durvalumab (MEDI4736)

F) Research Hypothesis: Is Durvalumab efficient in delay progression in patients with persistent disease after chemoradiation for locally advanced esophageal squamous cell carcinoma?

G) Objectives:

G1) Primary Objectives:

To assess the efficacy of durvalumab treatment in terms of 6-month progression-free survival.

G2) Secondary Objective(s):

To assess the incidence of grade 3 or higher toxicities; To further assess the efficacy of durvalumab in terms of overall survival, incidence of locoregional progression and incidence of distant progression.>>

G3) Exploratory Objective(s):

To investigate the relationship between immune biomarkers within the tumor microenvironment (immunohistochemistry) with efficacy outcomes with durvalumab

H) Study Design: Single arm phase II trial

I) Number of Centers: 1

J) Number of Patients:22

K) Study Population:

Patients with locally advanced unresectable or inoperable esophageal squamous cell carcinoma who had a persistent disease after completing definitive chemoradiotherapy, with no progressive disease.

L) Inclusion Criteria:

* Body weight >30kg and body mass index ≥ 16 kg / m2;
* Patients who are aphagic or able to ingest only liquids should also receive enteral nutritional support before inclusion in the study;
* Patients with histologically and/or cytologically confirmed esophageal or esophagogastric junction (Siewert I or II) squamous cell carcinoma, irrespective of PD-1/PD-L1 or any other biomarker expression;
* Patients who had a persistent disease 6-8 weeks after completing chemoradiotherapy with at least 50 Gy and platinum-based chemo and without clinical complete response or progressive disease;
* CT scans within 4 weeks revealing persistent disease;
* Must be included <12 weeks after completing chemoradiotherapy to ensure durvalumab begins no later than 16 weeks after completion of chemoradiotherapy;
* Patients unsuitable to salvage esophagectomy;
* All the tumor volume should have been treated with CRT (included in the radiation field); ECOG 0 - 1;
* Age 18 years or older;
* Life expectancy of higher than 3 months;
* Laboratory values must meet the following criteria: Absolute neutrophil count (ANC) > 1.5 (>1500 per mm3); Platelet count ≥ 100 x109/L. Hemoglobin >9.0 g/dL. Creatinine < 1.5 times institutional ULN or CrCl > 40 mL/min. AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal. Serum bilirubin ≤ 1.5 times institutional ULN (This will not apply to patients with confirmed Gilbert's syndrome - persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology, who will be allowed only in consultation with their physician)
* All toxicities attributed to prior chemoradiotherapy other than alopecia, fatigue, or peripheral neuropathy must have resolved to grade 2 or less.

M) Exclusion Criteria:

* Presence of any site of metastatic disease, including lymph node which has not been included in radiation field;
* Are currently receiving or have had prior use of immunosuppressive medication within 28 days before the first dose of study drug (10 milligrams/day of prednisone or an equivalent corticosteroid is allowed);
* Received any immunotherapy for esophageal cancer;
* Has known active hepatitis B, hepatitis C or human immunodeficiency virus (HIV1/2 antibodies);
* Has known active or prior autoimmune disease, except for:
* skin diseases (vitiligo, psoriasis, alopecia)
* diabetes mellitus type 1, with hormone replacement
* hypothyroidism, with hormone replacement
* Receipt of live attenuated vaccination within 30 days prior to study entry.
* Grade 3 or higher pulmonary toxicity of dyspnea, hypoxia, or pneumonitis experienced during chemoradiation;
* Presence of tracheoesophageal fistula that has not been treated with endoprosthesis>>

N) Investigational Product(s), Dose and Mode of Administration:

Patients in the durvalumab (MEDI4736) monotherapy treatment group will receive 1500 mg durvalumab (MEDI4736) via IV infusion Q4W <<for up to a maximum of 12 months (up to 13 doses/cycles) with the last administration on week 48 unless there is unacceptable toxicity, disease progression, withdrawal of consent, or another discontinuation criterion is met. If a patient's weight falls to 30 kg or below for 1 week or longer ( ≥ 7 days) durvalumab will be permanently discontinued.

O) Study Assessments and Criteria for Evaluation:

O.1) Safety Assessments:

Safety assessments will be performed in accordance with the National Cancer Institute Common Terminology Criteria, version 5.0.

At least every 4 weeks, during each visit, data on toxicity on treatment will be evaluated.

Laboratory analysis will also be performed at least every 4 weeks to assess toxicity.

O.2) Efficacy Assessments:

Patients will undergo tumor assessments with cross-sectional imaging at study site at start and then 8 ± 1w until complete 12 months after first dose; Patients who have disease control following completion of 12 months (13 cycles) of treatment will continue to have objective tumor assessment q12w ± 1w for more 12 months or until disease progression (whichever comes first); Patients who are withdrawn from durvalumab treatment for reasons other than confirmed PD (e.g toxicity) will continue to have objective tumor assessments q8w ± 1w until complete 12 months after first dose. Then, they will have objective tumor assessments q12w ± 1w for more 12 months (24 months after first dose) or until disease progression; Measurable target and nontarget lesions will be assessed according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).

P) Statistical Methods and Data Analysis:

Safety analysis will be performed considering all enrolled patients who received at least one dose of durvalumab; Efficacy analysis will be performed using intention-to-treat approach; Will be used an alpha error of 0.05 (1-sided) and a power (1 - beta error) of 90%; Primary endpoint will be 6-month progression free survival rate; Secondary endpoints will be overall survival, incidence of locoregional progression and incidence of distant progression; Locoregional progression is defined when an in-field lesion (primary tumor or lymph nodes) is the first site of progression or in case of worsening dysphagia with an upper endoscopy revealing an unequivocal local progression; Distant progression is defined when an out-field lesion (lymph node, visceral, bone) is the first site of progression; We estimate 12 months of recruitment, with 2 patients per month; Overall survival will be estimated using Kaplan-Meier method.

Q) Sample Size Determination:

Single arm phase II trial; Will be estimated p0 (null-hypothesis 6-month PFS) as 10%; Will be estimated p1 (alternative hypothesis 6-month PFS) as 35%; With an estimated dropout rate of 10%, our sample size will be 22 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Body weight >30kg and body mass index ≥ 16 kg / m2;
2. Patients aphagic or able to ingest only liquids should also receive enteral nutritional sup-port before being included in the study;
3. Patients must have histologically confirmed esophageal or esophagogastric junction (Siewert I or II) squamous cell carcinoma, irrespective of PD-1/PD-L1 or other biomarkers expression;
4. Patients must have had a persistent disease 6-8 weeks after completing chemoradiotherapy with at least 50 Gy and platinum-based chemo and without complete response or progressive disease, based on upper endoscopy and/or CT scans;
5. Patients must have realized CT scans within 6-8 weeks after completion of chemoradiotherapy, revealing persistent disease;
6. Patients must be included <12 weeks after completing chemoradiotherapy;
7. Patients must be unsuitable to salvage esophagectomy, according multidisciplinary local board;
8. All the tumor volume should have been treated with CRT (included in the radiation field);
9. Eastern Cooperative Oncology Group (ECOG)>><<World Health Organisation (WHO) performance status of 0 or 1;
10. Male or female aged 18 years or older at time of study entry;
11. Life expectancy of > 12 weeks;
12. Adequate normal organ and marrow function as defined below:

    * Haemoglobin ≥9.0 g/dL
    * Absolute neutrophil count (ANC) 1.5 x (> 1500 per mm3)
    * Platelet count ≥100 x 109/L
    * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). <<This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
    * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
    * Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance: CrCl, mL/min = (140 - age) × (weight, kg) × (0.85 if female) / (72 × Cr)
13. All toxicities attributed to prior chemoradiotherapy other than alopecia, fatigue, or peripheral neuropathy must have resolved to grade 2 or less;

Exclusion Criteria:

1. Patients with metastases including lymph node not included in the radiation field;
2. Patients currently receiving or have had prior use of immunosuppressive medication within 28 days before the first dose of study drug (10 milligrams/day of prednisone or an equivalent corticosteroid is allowed);
3. Received any immunotherapy for esophageal cancer;
4. Patients with active hepatitis B, hepatitis C or human immunodeficiency virus (HIV1/2 antibodies);
5. Has known active or prior autoimmune disease, except for:

   * skin diseases (vitiligo, psoriasis, alopecia)
   * diabetes mellitus type 1, with hormone replacement
   * hypothyroidism, with hormone replacement
6. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP.
7. Grade 3 or higher pulmonary toxicity of dyspnea, hypoxia, or pneumonitis experienced during chemoradiation;
8. Presence of fistula between esophagus and trachea unless treated with endoscopic prosthesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Six-month progression-free survival | 6 months
  The primary endpoint is the percentage of subjects who remain progression free at 6 months using investigator assessments according to RECIST 1.1

SECONDARY OUTCOMES:
Incidence of Treatment-Related Adverse Events [Safety and Tolerability] | From time of informed consent through treatment period (12 months) or up to 12 months post last dose of study treatment.
  Incidence of grade 3 or higher toxicities graded according to NCI CTCAE (version 5.0)
Overall survival | From time of informed consent until the date of death from any cause, assessed up to 60 months
  Time from randomization until death from any cause.
Incidence of locoregional progression | From time of informed consent through treatment period (12 months) or up to 12 months post last dose of study treatment.
  Defined as the number of patients whose the first site of progression was in field.
Incidence of distant progression | From time of informed consent through treatment period (12 months) or up to 12 months post last dose of study treatment.
  Defined as the number of patients whose the first site of progression was distant.

OTHER OUTCOMES:
Six-month progression-free survival according to immune biomarkers | 6 months
  Percentage of subjects who remain progression free at 6 months according to immune-related or response-related markers by immunohistochemistry (PD-1, PD-L1, CTLA-4, CD3, CD4, CD8, CD45RO, forkhead box P3, granzyme B, OX40, cleaved caspase 3 and Ki67).

CONTACTS AND LOCATIONS:
Overall Officials: Tiago B de Castria, MD PhD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Instituto do Câncer do Estado de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No